CLINICAL TRIAL: NCT01367639
Title: Pilot Randomized Controlled Trial of Inquiry Based Stress Reduction (IBSR) Program for BRCA1/2 Mutation Carriers
Brief Title: Trial of Inquiry Based Stress Reduction (IBSR) Program for BRCA1/2 Mutation Carriers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-8400-EF-CTIL
Record Dates: First submitted 2011-05-31; First posted 2011-06-07 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
Keywords: BRCA 1/2 Carriers; IBSR; The Work; Randomized clinical trial
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): Inquiry Based Stress Reduction (IBSR) program
  Interventions: Behavioral: Inquiry Based Stress Reduction (IBSR) program

INTERVENTIONS:
Behavioral: Inquiry Based Stress Reduction (IBSR) program — The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie, trains participants to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and provides skills for self-inquiry and management of stressful thoughts that can be easily implemented in daily life

SUMMARY:
Breast cancer (BC) is a major health problem and the most prevalent cancer among women.In a substantial proportion of familial cases, germ-line mutations in either BRCA1/2 can be detected. The only proven modality for active risk reduction (rather than passive early detection), is prophylactic surgery - prophylactic mastectomy and oophorectomy. While the majority of Jewish mutation carriers elect to undergo prophylactic oophorectomy at about age 40 years, in Israel only a minority perform prophylactic mastectomy. Another ramification of being a mutation carrier is the emotional stress associated with that discovery.Genetic information has profound implications for mutation carriers. The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie, trains participants to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and provides skills for self-inquiry and management of stressful thoughts that can be easily implemented in daily life [ ]. Therefore, on the basis of previous data and beneficial observations we postulate that the clinical utility of IBSR mediation program may improve psychological and physical symptoms and quality of life among asymptomatic (oncologically healthy) BRCA1/ BRCA2 mutation carriers. Thus, we will conduct a pilot randomized controlled trial to scientifically investigate the effect of this intervention effects on BRCA1/2 mutation carriers.

DETAILED DESCRIPTION:
Main Goals: To investigate whether IBSR intervention is efficacious in improving quality of life, psychological and physical status in BRCA1/2 mutation carriers.

Secondary-goal: To Assess feasibility of IBSR intervention by examining attendance, drop-out rates, and program satisfaction.

Hypothesis Participants' ability to deal with emotional difficulties will be improved following participation in the IBSR intervention. This will be reflected in improving the values of psychological measures, such as quality of sleep, cancer related worry, family support, depression and anxiety, after the intervention (among participants in the intervention group, but not in the control group).

Study population: Eligible individuals are women who are carriers of one of the predominant Jewish mutations in BRCA1/2 genes at the Meirav Center, Sheba Medical center over the past 10 years. All eligible women will be contacted by the staff of the Meirav Center and will be offered participation during routine follow up visits at the high risk clinic, by phone or a letter. Interested individuals will be scheduled to attend a meeting at a time of their convenience with the PI or the Co PIs to explain the study aims and goals. After the participant has agreed and signed the informed consent she is considered eligible.

ELIGIBILITY:
Inclusion Criteria:

* Women who are carriers of one of the predominant Jewish mutations in BRCA1/2 genes, age 35 years or older, with no current or past history of cancer (except BCC), who are willing to sign an informed consent, and present mental clarity by the ability to comprehend and fulfill all the questionnaires.

Exclusion Criteria:

* Diagnosed with breast or ovarian cancer or any other cancer, self reported Pregnancy, risk reduction mastectomy, severe psychiatric diagnosis (e.g. bipolar disorder).

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
global psychology functioning(GSI) | 12 Weeks
Sleep quality (PSQI) | 12 weeks

SECONDARY OUTCOMES:
Family support PSS-Fa | 12 weeks
cancer related worry (CRW) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Friedman, Prof., Principal Investigator — Sheba Medical Center; Shahar Lev-ari, Dr., Study Director — Department of health promotion, faculty of medicine, Tel Aviv University
Locations (1):
- Sheba Medical Center, Tel Aviv, Israel